CLINICAL TRIAL: NCT02650674
Title: Determination of the Glycaemic Index and Insulinaemic Index Values of Five Cereal Products
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mondelēz International, Inc. (Industry)
Collaborators: University of Sydney (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: KBE043
Record Dates: First submitted 2015-10-30; First posted 2016-01-08 (Estimated); Last update posted 2017-09-14 (Actual); Status verified 2017-09

CONDITIONS: Metabolic Disorder
Keywords: glycemic & insulin response; SDS; cereal product; Nutrition; Carbohydrate; Absorption; Intestine
MeSH Terms: conditions — Metabolic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Product A: NP-0148 (Experimental): Cereal product belVita Milk & Cereals - High in SDS
  Interventions: Other: Product A: NP-0148
- Product B: NP-0149 (Experimental): Cereal product belVita Honey & Nuts - High in SDS
  Interventions: Other: Product B: NP-0149
- Product C: NP-0150 (Experimental): Cereal product belVita Mixed Berry - High in SDS
  Interventions: Other: Product C: NP-0150
- Product D: NP-0151 (Experimental): Cereal product Kellogg's Corn Flakes - Low in SDS - Low in fat
  Interventions: Other: Product D: NP-0151
- Product E: NP-0152 (Experimental): Cereal product Kellogg's Trésor Duo Choco - Low in SDS
  Interventions: Other: Product E: NP-0152
- Glucose reference (Experimental): Glucose solution performed on three occasions
  Interventions: Other: Glucose solution

INTERVENTIONS:
Other: Product A: NP-0148 — Portions of cereal product calculated to provide 50 g of available carbohydrates will be served with 250 mL water.
  Arms: Product A: NP-0148
Other: Glucose solution — Glucose solution providing 50 g of available carbohydrates in 250 ml of water. This will be performed 3 times
  Arms: Glucose reference
Other: Product B: NP-0149 — Portions of cereal product calculated to provide 50 g of available carbohydrates will be served with 250 mL water.
  Arms: Product B: NP-0149
Other: Product C: NP-0150 — Portions of cereal product calculated to provide 50 g of available carbohydrates will be served with 250 mL water.
  Arms: Product C: NP-0150
Other: Product D: NP-0151 — Portions of cereal product calculated to provide 50 g of available carbohydrates will be served with 250 mL water.
  Arms: Product D: NP-0151
Other: Product E: NP-0152 — Portions of cereal product calculated to provide 50 g of available carbohydrates will be served with 250 mL water.
  Arms: Product E: NP-0152

SUMMARY:
This study aimed at determining the Glycaemic Index and Insulinaemic Index Values of Five Cereal Products in two different ethnic groups.

DETAILED DESCRIPTION:
This study aimed at determining the Glycaemic Index and Insulinaemic Index Values of Five Cereal Products in two different ethnic groups. It is a laboratory-based research study, conducted in two different ethnic groups, with an open cross-over design, including 24 healthy non-smoking voluntary subjects, aged from 18 to 45 years. 12 subjects will be Caucasian and 12 subjects will be Asian. 8 test sessions per subject are included in the study. Foods are consumed in a random order according to a randomisation list. The impact of the ethnic group and the products will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18-45 years.
* Non-smoker.
* BMI values: between 19-25 kg/m2 (bounds included) for Caucasian subjects and between 19-23 kg/m2 (bounds included) for Asian subjects (WHO expert consultation).
* Ethnicity: Caucasian subjects will have both parents from Caucasian ancestry. Asian subjects will have both parents from Asian country and will be born in an Asian country. Asian countries are: Brunei Darussalam, Cambodia, China, Dem. People's Republic of Korea, Hong Kong SAR (China), Indonesia, Japan, Lao People's Democratic Republic, Macao SAR (China), Malaysia, Mongolia, Myanmar, Philippines, Republic of Korea, Singapore, Taiwan, Thailand, Viet Nam.
* Sex ratio: Around half of the subjects should be male and half of the subjects should be female within each study group. A plus or minus 1 subject tolerance will be accepted.
* Healthy subjects with:

Normal glucose tolerance Normal laboratory values for various measures of metabolic health (full blood count, gamma-GT, AST, ALT, glucose, TAGs, total cholesterol, HDL-cholesterol, LDL-cholesterol); Normal systolic blood pressure (100-150 mmHg); Normal diastolic blood pressure (60-90 mmHg); Normal resting heart rate (50-90 beats per minutes after 3 minutes rest).

* Stable dietary habits; normal eating patterns; no history of eating disorders or strict dieting.
* Moderate level of physical activity (from basic daily activity to a high level of physical activity (regular physical activity at least 3 times per week))
* Able to fast for at least 10 hours the night before each test session.
* Able to refrain from eating legumes and drinking alcohol the day before each test session.
* Subject covered by social security or covered by a similar system
* Subject not taking any treatment for anorexia, weight loss, or any form of treatment likely to interfere with metabolism or dietary habits
* Subject having given written consent to take part in the study.

Exclusion Criteria:

* Following a restrictive diet.
* Family history of Diabetes Mellitus or obesity
* Suffering from any clinical, physical or mental illness.
* Suffering from any food allergies or hypersensitivities (wheat, milk, egg, nuts, etc).
* Taking any regular prescription medication at the time of inclusion (except regular oral contraception medication)
* Female who is pregnant (positive test results), lactating, planning pregnancy or not using acceptable contraceptive.
* Females who consistently suffer from premenstrual tension and marked changes in appetite during their menstrual cycle.
* Subject having taken part in another clinical trial within the last week.
* Subject currently taking part in another clinical trial or being in the exclusion period of another clinical trial.
* Subject undergoing general anaesthesia in the month prior to inclusion.
* Subject in a situation which in the investigator's opinion could interfere with optimal participation in the present study or could constitute a special risk for the subject.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2015-10; Primary Completion 2016-03 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Glycaemic index values of five cereal products | 2 hours after food consumption
  Determination of GI in both Caucasian and Asian subjects

SECONDARY OUTCOMES:
Glycaemic response assessed by the glycemic index (GI) values of five cereal products | 2 hours after food consumption
  Determination of GI in the global population
Glycaemic response assessed by the postprandial changes in glycaemia over 2 hours (iAUC0-120) after consumption of the test products | 2 hours after food consumption
  This parameter will be analyzed first in both Caucasian and Asian populations and second globally
Glycaemic response assessed by the kinetic of glycemia over the 120 minutes | 2 hours after food consumption
  This parameter will be analyzed first in both Caucasian and Asian populations and second globally
Glycaemic response assessed by the peak value of glycemia | 2 hours after food consumption
  This parameter will be analyzed first in both Caucasian and Asian populations and second globally
Glycaemic response assessed by the delta value between baseline and peak values of glycemia | 2 hours after food consumption
  This parameter will be analyzed first in both Caucasian and Asian populations and second globally
Insulinaemic response assessed by the insulinemic index (II) values of five cereal products | 2 hours after food consumption
  This parameter will be analyzed first in both Caucasian and Asian populations and second globally
Insulinaemic response assessed by the postprandial changes in insulinemia over 2 hours (iAUC0-120) after consumption of the test products | 2 hours after food consumption
  This parameter will be analyzed first in both Caucasian and Asian populations and second globally
Insulinaemic response assessed by the kinetic of insulinemia over the 120 minutes | 2 hours after food consumption
  This parameter will be analyzed first in both Caucasian and Asian populations and second globally
Insulinaemic response assessed by the peak value of insulinemia | 2 hours after food consumption
  This parameter will be analyzed first in both Caucasian and Asian populations and second globally
Insulinaemic response assessed by the delta value between baseline and peak values of insulinemia | 2 hours after food consumption
  This parameter will be analyzed first in both Caucasian and Asian populations and second globally
Insulin / glucose ratio (II/GI) evaluation of five cereal products | 2 hours after food consumption
  This parameter will be analyzed first in both Caucasian and Asian populations and second globally
Postprandial changes in insulin / glucose over 2 hours (iAUC0-120) after consumption of the test products | 2 hours after food consumption
  This parameter will be analyzed first in both Caucasian and Asian populations and second globally
Kinetic of insulin / glucose over the 120 minutes | 2 hours after food consumption
  This parameter will be analyzed first in both Caucasian and Asian populations and second globally
Peak value of insulin / glucose ratio | 2 hours after food consumption
  This parameter will be analyzed first in both Caucasian and Asian populations and second globally
Delta peak value between baseline and peak values of insulin / glucose ratio | 2 hours after food consumption
  This parameter will be analyzed first in both Caucasian and Asian populations and second globally

CONTACTS AND LOCATIONS:
Overall Officials: Jennie Brand Miller, Principal Investigator — University of Sydney
Locations (1):
- University of Sydney, Sydney, New South Wales, Australia